CLINICAL TRIAL: NCT00931632
Title: Inhaled Nitric Oxide (INO) for the Prevention of Bronchopulmonary Dysplasia (BPD) in Preterm Infants Requiring Mechanical Ventilation or Positive Pressure Support on Days 5-14 After Birth
Brief Title: Inhaled Nitric Oxide (INO) for the Prevention of Bronchopulmonary Dysplasia (BPD) in Preterm Infants
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Mallinckrodt (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Triple | Purpose: Treatment
Other Study IDs: IK-3001-BPD-301
Record Dates: First submitted 2009-07-01; First posted 2009-07-02 (Estimated); Results first posted 2015-08-11 (Estimated); Last update posted 2017-12-04 (Actual); Status verified 2017-10

CONDITIONS: Bronchopulmonary Dysplasia
Keywords: Bronchopulmonary Dysplasia, BPD
MeSH Terms: conditions — Bronchopulmonary Dysplasia | interventions — Endothelium-Dependent Relaxing Factors; Nitrogen

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Inhaled Nitric Oxide (Experimental): Inhaled Nitric Oxide
  Interventions: Drug: Inhaled Nitric Oxide
- Placebo (Placebo Comparator): Nitrogen Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Inhaled Nitric Oxide — Inhaled Nitric Oxide will be administered continuously starting at 20ppm into the inspiratory limb of the ventilator circuit in mechanically ventilated subject using an INOvent delivery system of by nasal cannula as needed for 24 days of therapy.
  Other Names: INOmax
  Arms: Inhaled Nitric Oxide
Drug: Placebo — Nitrogen gas will be administered in the same manner as the experimental drug.
  Other Names: Nitrogen gas
  Arms: Placebo

SUMMARY:
This phase 3, multi-center, double blind, placebo-controlled, randomized clinical trial will attempt to demonstrate if preterm infants who require mechanical ventilation and/or positive pressure support at any point during days 5 to 14 after birth may benefit from treatment with iNO.

DETAILED DESCRIPTION:
Multi-center, double blind, placebo-controlled, randomized clinical trial. Infants who meet all enrollment criteria at any point during days 5 to 14 after birth will be randomized to inhaled NO starting at 20 ppm, or matching placebo, by means of a blinded INOvent® delivery device. All infants will receive 24 days of therapy, following a dose reduction schedule. Infants who are extubated before 24 days will continue therapy via nasal continuous positive airway pressure (CPAP) or nasal cannula to complete 24 days' of therapy. The primary outcome measure will be survival without BPD at 36 weeks gestational age using a physiologic assessment of BPD.

ELIGIBILITY:
Inclusion Criteria:

* Preterm infants who are:

  1. 500 to 1250 grams at birth
  2. < 30 weeks gestational age
  3. 5 to 14 days of age (inclusive) at the time of entry
  4. Requiring mechanical ventilation or for those infants ≤ 800 grams, positive pressure support (including CPAP) for respiratory insufficiency on days 5 to 14 days of age (inclusive)

Exclusion Criteria:

1. Preterm infants with life-threatening anomalies (cranial, cardiac, thoracic, chromosomal) or congenital diaphragmatic hernia with lung hypoplasia, or any subject who will not receive complete intensive care
2. Preterm infants with bilateral Grade 4 intraventricular hemorrhage (IVH)
3. Subjects who are dependent on right to left shunting to maintain the systemic circulation
4. Preterm infants who received prior iNO therapy
5. Use of another investigational agent

Ages: 5 Days to 14 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 451 (Actual)
Dates: Start 2009-11; Primary Completion 2013-05 (Actual); Study Completion 2014-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: James Baldassarre, MD, Study Director — Mallinckrodt
Locations (33):
- United States (31):
  - Phoenix Children's Hospital, Phoenix, Arizona
  - St. Joseph's Hospital and Medical Center, Phoenix, Arizona
  - Loma Linda University School of Medicine, Loma Linda, California
  - Children's Hospital of Orange County, Orange, California
  - Stanford University School of Medicine, Palo Alto, California
  - Rady Children's Hospital of San Diego, San Diego, California
  - Sharp Mary Birch Hospital for Women and Newborns, San Diego, California
  - Connecticut Children's Medical Center, Hartford, Connecticut
  - Winnie Palmer Hospital for Women and Babies, Orlando, Florida
  - University of So Florida College of Medicine, Tampa, Florida
  - Medical College of Georgia, Augusta, Georgia
  - Advocate Lutheran General Children's Hospital, Park Ridge, Illinois
  - Riley Hospital for Children, Indianapolis, Indiana
  - University of Louisville School of Medicine, Louisville, Kentucky
  - Hennepin County Medical Center, Minneapolis, Minnesota
  - Saint Barnabas Medical Center, Livingston, New Jersey
  - Jersey Shore University Medical Center, Neptune City, New Jersey
  - Robert Wood Johnson University Hospital, New Brunswick, New Jersey
  - Winthrop University Hospital, Mineola, New York
  - Montefiore Medical Center, The Bronx, New York
  - Maria Fareri Children's Hospital at Westchester Medical Center, Valhalla, New York
  - WakeMed Faculty Physicians, Neonatology, Raleigh, North Carolina
  - Mercy Children's Hospital, Toledo, Ohio
  - Saint Francis Children's Hospital, Tulsa, Oklahoma
  - Greenville Memorial Hospital, Greenville, South Carolina
  - Sanford Children's Hospital, Sioux Falls, South Dakota
  - Cook Children's Medical Center, Fort Worth, Texas
  - Primary Children's Medical Center, Salt Lake City, Utah
  - Virginia Commonwealth University, Richmond, Virginia
  - Wheaton Franciscan Healthcare, Milwaukee, Wisconsin
  - Children's Corporate Center, Division of Neonatology, Wauwatosa, Wisconsin
- Canada (2):
  - University of Calgary, Calgary, Alberta
  - Centre Hospitalier Universitaire de Quebec, Québec

REFERENCES:
- [Result] Hasan SU, Potenziano J, Konduri GG, Perez JA, Van Meurs KP, Walker MW, Yoder BA; Newborns Treated With Nitric Oxide (NEWNO) Trial Group. Effect of Inhaled Nitric Oxide on Survival Without Bronchopulmonary Dysplasia in Preterm Infants: A Randomized Clinical Trial. JAMA Pediatr. 2017 Nov 1;171(11):1081-1089. doi: 10.1001/jamapediatrics.2017.2618. PMID 28973344
- See also: Related Info — http://jamanetwork.com/journals/jamapediatrics/article-abstract/2654598

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Inhaled Nitric Oxide | Placebo
Started | 229 (Randomized) | 222 (Randomized)
Completed | 208 (Completed at 36 weeks Postmenstrual Age (PMA)) | 204 (Completed at 36 weeks Postmenstrual Age (PMA))
Not Completed | 21 | 18
Not completed — Withdrawal by Subject | 2 | 3
Not completed — Adverse Event | 19 | 15

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Inhaled Nitric Oxide | Placebo | Total
Number analyzed (Participants) | 229 | 222 | 451
Age, Customized [Number; unit: participants] — Preterm infants < 30 weeks Gestational Age (GA)
  participants | 229 | 222 | 451
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 114 | 106 | 220
  Male | 115 | 116 | 231
Race/Ethnicity, Customized [Number; unit: participants]
  White | 120 | 85 | 205
  Black | 55 | 62 | 117
  Hispanic | 40 | 48 | 88
  American Indian | 1 | 12 | 13
  Asian | 1 | 5 | 6
  Pacific Islander | 1 | 0 | 1
  Other | 11 | 10 | 21
Region of Enrollment [Number; unit: participants]
  United States | 209 | 203 | 412
  Canada | 20 | 19 | 39

OUTCOME MEASURES:

1. Primary Outcome: Survival Without BPD at 36 Weeks
Time Frame: Baseline, 36 weeks PMA
Population: Subjects with missing primary outcome or who crossed over to open-label iNO during the blinded treatment period were considered as failures
Measure: Number; unit: participants
Arm/Group | Inhaled Nitric Oxide | Placebo
Number analyzed (Participants) | 229 | 222
participants
  Alive without BPD at 36 weeks GA | 80 | 70
  Death or had BPD at 36 weeks GA | 149 | 152
Statistical Analysis 1: Comparison: Inhaled Nitric Oxide vs Placebo; Test type: Superiority or Other; p = 0.427, Mantel Haenszel

2. Secondary Outcome: Days of Airway Pressure Support - Intent-to-treat Population
Description: Airway pressure support includes conventional mechanical ventilation, conventional, high frequency oscillatory ventilation, jet, continuous positive airway pressure, and other.
Time Frame: Through hospital discharge, an average of 105 days for placebo and 108 days for INO
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Inhaled Nitric Oxide | Placebo
Number analyzed (Participants) | 229 | 220
Days | 53.7 (42.16) | 55.3 (40.45)

3. Secondary Outcome: Length of Birth Hospitalization
Time Frame: Through hospital discharge, an average of 105 days for placebo and 108 days for INO
Population: Number of subjects within the Intent-to-treat population with available data
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Inhaled Nitric Oxide | Placebo
Number analyzed (Participants) | 201 | 203
Days | 108.3 (54.03) | 105.0 (36.69)

4. Secondary Outcome: Number and Percentage of Participants With Use of Postnatal Corticosteroids for Bronchopulmonary Dysplasia
Time Frame: Through hospital discharge, an average of 105 days for placebo and 108 days for INO
Population: Intent-to-treat population
Measure: Count of Participants; unit: Participants
Arm/Group | Inhaled Nitric Oxide | Placebo
Number analyzed (Participants) | 229 | 222
Participants
  Yes | 95 | 91
  No | 134 | 131

5. Secondary Outcome: Number and Percentage of Participants With Use of Postnatal Corticosteroids for Any Medical Reason
Time Frame: Through hospital discharge, an average of 105 days for placebo and 108 days for INO
Population: Intent-to-treat population
Measure: Count of Participants; unit: Participants
Arm/Group | Inhaled Nitric Oxide | Placebo
Number analyzed (Participants) | 229 | 222
Participants | 154 | 145

6. Secondary Outcome: Systemic Use of Postnatal Corticosteroids for Any Medical Reason
Time Frame: Through hospital discharge, an average of 105 days for placebo and 108 days for INO
Population: Intent-to-treat population
Measure: Count of Participants; unit: Participants
Arm/Group | Inhaled Nitric Oxide | Placebo
Number analyzed (Participants) | 229 | 222
Participants | 144 | 131

7. Secondary Outcome: Number of Days of Oxygen Use
Time Frame: Through hospital discharge, an average of 105 days for placebo and 108 days for INO
Population: Number of subjects within the Intent-to-treat population with available data
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Inhaled Nitric Oxide | Placebo
Number analyzed (Participants) | 207 | 212
Days | 91.0 (59.26) | 88.0 (40.91)

8. Secondary Outcome: Severity of Bronchopulmonary Dysplasia
Description: Severity of bronchopulmonary dysplasia defined by the fraction of inspired O2 concentration (FiO2) requirement.
Time Frame: 36 weeks
Population: Number of subjects within the Intent-to-treat population with available data
Measure: Count of Participants; unit: Participants
Arm/Group | Inhaled Nitric Oxide | Placebo
Number analyzed (Participants) | 207 | 211
Participants
  0 = None | 1 | 2
  1 = Mild | 80 | 72
  2 = Moderate | 83 | 82
  3 = Severe | 43 | 55

ADVERSE EVENTS:
Time Frame: Through treatment completion, up to 24 days
Description: During treatment of 24 day course
Arm/Group | Inhaled Nitric Oxide | Placebo
All-Cause Mortality (participants affected / at risk) | 12/229 | 8/220
Serious Adverse Events (participants affected / at risk) | 105/229 | 100/220
Other Adverse Events (participants affected / at risk) | 169/229 | 143/220
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Inhaled Nitric Oxide (N=229) | Placebo (N=220)
Patent ductus arteriosus (Congenital, familial and genetic disorders) | 34 | 34
Necrotising enterocolitis neonatal (Gastrointestinal disorders) | 11 | 15
Sepsis (Infections and infestations) | 25 | 27
Anemia neonatal (Blood and lymphatic system disorders) | 4 | 6
Thrombocytopenia (Blood and lymphatic system disorders) | 2 | 4
Hemolytic anemia (Blood and lymphatic system disorders) | 0 | 1
Neutropenia (Blood and lymphatic system disorders) | 0 | 1
Bradycardia (Cardiac disorders) | 1 | 0
Cardio-respiratory arrest (Cardiac disorders) | 1 | 1
Cardiopulmonary failure (Cardiac disorders) | 1 | 0
Pneumopericardium (Cardiac disorders) | 1 | 0
Supraventricular tachycardia (Cardiac disorders) | 1 | 0
Ventricular fibrillation (Cardiac disorders) | 1 | 0
Atrial thrombosis (Cardiac disorders) | 0 | 1
Cardiac arrest (Cardiac disorders) | 0 | 1
Persistent fetal circulation (Congenital, familial and genetic disorders) | 1 | 2
Adrenogenital syndrome (Congenital, familial and genetic disorders) | 0 | 1
Hereditary spherocytosis (Congenital, familial and genetic disorders) | 0 | 1
Intestinal perforation (Gastrointestinal disorders) | 8 | 4
Abdominal distension (Gastrointestinal disorders) | 2 | 1
Gastrointestinal perforation (Gastrointestinal disorders) | 1 | 1
Inguinal hernia (Gastrointestinal disorders) | 1 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 1 | 0
Ileal perforation (Gastrointestinal disorders) | 0 | 1
Intestinal obstruction (Gastrointestinal disorders) | 0 | 1
Esophageal perforation (Gastrointestinal disorders) | 0 | 1
Hepatic function abnormal (Hepatobiliary disorders) | 0 | 1
Pneumoperitoneum (Gastrointestinal disorders) | 0 | 1
Hyperbilirubinemia (Hepatobiliary disorders) | 0 | 1
Staphylococcal sepsis (Infections and infestations) | 7 | 4
Group B streptococcus neonatal sepsis (Infections and infestations) | 3 | 0
Pneumonia (Infections and infestations) | 3 | 7
Septic shock (Infections and infestations) | 3 | 1
Fungal sepsis (Infections and infestations) | 2 | 0
Pneumonia bacterial (Infections and infestations) | 2 | 2
Urinary tract infection (Infections and infestations) | 2 | 2
Bacterial sepsis (Infections and infestations) | 1 | 2
Beta hemolytic streptococcal infection (Infections and infestations) | 1 | 0
Enterococcal sepsis (Infections and infestations) | 1 | 0
Lung infection pseudomonal (Infections and infestations) | 1 | 0
Pneumonia staphylococcal (Infections and infestations) | 1 | 2
Staphylococcal bacteremia (Infections and infestations) | 1 | 0
Staphylococcal infection (Infections and infestations) | 1 | 0
Abdominal abscess (Infections and infestations) | 0 | 1
Enterobacter sepsis (Infections and infestations) | 0 | 2
Klebsiella sepsis (Infections and infestations) | 0 | 1
Lung abscess (Infections and infestations) | 0 | 1
Meningitis candida (Infections and infestations) | 0 | 1
Streptococcal sepsis (Infections and infestations) | 0 | 1
Tracheitis (Infections and infestations) | 0 | 1
Urinary tract infection fungal (Infections and infestations) | 0 | 1
Bacterial test positive (Investigations) | 1 | 0
CST culture positive (Investigations) | 1 | 1
Candida test positive (Investigations) | 0 | 1
Hyperkalemia (Metabolism and nutrition disorders) | 1 | 0
Metabolic acidosis (Metabolism and nutrition disorders) | 1 | 3
Hydrocephalus (Nervous system disorders) | 3 | 2
Intraventricular hemorrhage neonatal (Nervous system disorders) | 3 | 3
Cerebral ventricle dilatation (Nervous system disorders) | 1 | 0
Encephalomalacia (Nervous system disorders) | 1 | 0
Hemorrhage intracranial (Nervous system disorders) | 1 | 0
Periventricular leukomalacia (Nervous system disorders) | 1 | 1
Renal failure (Renal and urinary disorders) | 1 | 1
Renal failure acute (Renal and urinary disorders) | 1 | 2
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 4 | 5
Infantile apnoeic attack (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Neonatal respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 3
Pulmonary hemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Emphysema (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pneumomediastinum (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Skin disorder (Skin and subcutaneous tissue disorders) | 0 | 1
Skin ulcer (Skin and subcutaneous tissue disorders) | 0 | 1
Thoracotomy (Surgical and medical procedures) | 0 | 1
Hypotension (Vascular disorders) | 7 | 2
Aortic thrombosis (Vascular disorders) | 1 | 0
Arterial spasm (Vascular disorders) | 1 | 0
Hypoperfusion (Vascular disorders) | 0 | 1
Thrombosis (Vascular disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Inhaled Nitric Oxide (N=229) | Placebo (N=220)
Hyponatraemia (Metabolism and nutrition disorders) | 66 | 50
Metabolic acidosis (Metabolism and nutrition disorders) | 29 | 29
Hyperglycemia (Metabolism and nutrition disorders) | 13 | 8
Feeding disorder neonatal (Metabolism and nutrition disorders) | 10 | 12
Bronchopulmonary dysplasia (Respiratory, thoracic and mediastinal disorders) | 29 | 21
Pulmonary edema (Respiratory, thoracic and mediastinal disorders) | 12 | 12
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 10 | 11

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Site shall use Confidential Information solely for the purposes of preforming its obligations under the Clinical Study Agreement and shall not, without Sponsor's prior written consent, publish, disseminate or otherwise disclose to any third party (including any of its affiliates) any Confidential Information. These obligations shall survive and continue for ten years after the termination or expiration of the Agreement or such longer period as required by Applicable Law.